CLINICAL TRIAL: NCT01992939
Title: The Effect of Heat on Blood and Oxygen Flow Readings Part 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Pittsburgh Healthcare System (U.S. Federal Agency)
Collaborators: Medline Industries (Industry)
Responsible Party: Principal Investigator, Cathy Abee, Medical Instrument Technologist, VA Pittsburgh Healthcare System
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PulsOx-002
Record Dates: First submitted 2013-11-13; First posted 2013-11-25 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-02

CONDITIONS: Healthy; Peripheral Vascular Disease; Vasoconstriction
Keywords: pulse; heat; blood circulation
MeSH Terms: conditions — Peripheral Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Non-Healthy Subjects arm (Active Comparator): Subjects in this arm will have peripheral vascular disease (PVD), vasoconstriction, or hypothermic extremities and they will receive two pulse oximetry probes. One probe will be a standard of care pulse oximetry probe and the second probe is the specialized pulse oximetry probe with external heat pack
  Interventions: Other: Specialized pulse oximetry probe with external heat pack; Other: Standard of Care Pulse Oximetry Probe
- Healthy Subjects Arm (Active Comparator): Subjects who do not have peripheral vascular disease (PVD), vasoconstriction, or hypothermic extremities will be considered healthy subjects and they will receive two pulse oximetry probes. One probe will be a standard of care pulse oximetry probe and the second probe is the specialized pulse oximetry probe with external heat pack.
  Interventions: Other: Specialized pulse oximetry probe with external heat pack; Other: Standard of Care Pulse Oximetry Probe

INTERVENTIONS:
Other: Specialized pulse oximetry probe with external heat pack — Pulse oximetry will be obtained using the specialized pulse oximetry probe with external heat pack for 45 minutes.
Other: Standard of Care Pulse Oximetry Probe — Pulse oximetry will be obtained using a standard of care pulse oximetry probe for 45 minutes.

SUMMARY:
This is the second part of a research study in order to determine if using a specialized pulse oximetry probe with external heat pack will help obtain oxygen saturation (SaO2) and heart rate (HR) during monitoring for patients with peripheral vascular disease (PVD), vasoconstriction, and hypothermic extremities. The inability to obtain accurate SaO2 and pulse readings can lead to misdiagnosis, incorrect treatment, or procedures to be canceled. SaO2 and pulse readings are important to maintain patient stability during diagnostic testing, surgical procedures and monitoring while in critical care areas. Changes in SaO2 and pulse are important to monitor in order to be able to compensate for any decrease in patient oxygen saturations during hemodynamic monitoring.

The primary aim of this study is to determine if using a specialized pulse oximetry probe with external heat pack will improve oxygenation readings in order to obtain SaO2 and pulse readings in patients with PVD, vasoconstriction, and hypothermic extremities as compared to readings obtained from an arterial blood gas.

The hypothesis is using a specialized pulse oximetry probe with external heat pack will help obtain more accurate pulse oximetry readings consistent with values obtained with an arterial blood gas.

DETAILED DESCRIPTION:
150 patients will be approached in order to ensure 110 patients will be enrolled in this study total. 30 patients will have peripheral vascular disease (PVD), vasoconstriction, or hypothermic extremities and 80 patients with no blood flow issues will be enrolled. The patients will serve as their own controls. Each patient will have a specialized pulse oximetry probe with external heat pack added to their extremity while measuring pulse oximetry. These SaO2 readings will be compared to SaO2 readings obtained from an arterial blood gas obtained during the course of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Able to give informed consent
3. Patients must be able to read and understand English.
4. Patients scheduled to enter the VA Pittsburgh Healthcare System catheterization lab

Arm 2 of the study:

1. The PI will determine if patients have poor circulation due to obstruction of the large arteries in their arms and legs (peripheral vascular disease (PVD), narrowing of their blood vessels (vasoconstriction), or extremities (arms, legs, etc) that are at least 3 degrees Fahrenheit below their normal body temperature. If patients do have any of the following they will be considered for arm 2. If they do not they will be considered for arm 1.

Exclusion Criteria:

In addition to the exclusions mentioned above, patients with the following conditions will be excluded from the trial:

1. Inability or unwillingness to sign informed consent with free will and sound mind, as determined by a score of <11 on the Evaluation to Sign Consent Form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2013-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Pulse Oximetry | measured at least every 5 minutes - day 1

SECONDARY OUTCOMES:
Arterial Blood Gas | measured once - day 1

OTHER OUTCOMES:
Temperature | measured at least every 5 minutes - day 1

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Abee, CRT, Principal Investigator — VA Pittsburgh Healthcare System
Locations (1):
- VA Pittsburgh Healthcare System, Pittsburgh, Pennsylvania, United States